CLINICAL TRIAL: NCT05101213
Title: Study Assessing the Feasibility, Safety and Efficacy of Genetically Engineered Glucocorticoid Receptor Knock Out Virus Specific CTL Lines for Viral Infections in Immunosuppressed Cancer Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0332; NCI-2021-09078 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0332 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-08-30; First posted 2021-11-01 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Adenovirus Infection; BK Virus Infection; Cytomegaloviral Infection; Hematopoietic and Lymphoid Cell Neoplasm; JC Virus Infection; Malignant Solid Neoplasm; Symptomatic COVID-19 Infection Laboratory-Confirmed
MeSH Terms: conditions — Adenoviridae Infections; Cytomegalovirus Infections; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment for viral infections (virus-specific CTLs) (Experimental): Patients receive virus-specific CTLs intravenously (IV) over 30 minutes. Patients with partial response, stable disease, or progressive disease may receive up to 8 additional infusions of virus-specific CTL at least 2 weeks between each infusion.
  Interventions: Biological: Virus-specific Cytotoxic T-lymphocytes

INTERVENTIONS:
Biological: Virus-specific Cytotoxic T-lymphocytes — Given IV
  Other Names: Virus-specific CTLs

SUMMARY:
This phase I trial tests the feasibility and safety of genetically modified cytotoxic T-lymphocytes in controlling infections caused by adenovirus (ADV), BK virus (BKV), cytomegalovirus (CMV), JC virus (JCV), or COVID-19 in immunocompromised patients with cancer. Viral infections are a leading cause of morbidity and mortality after hematopoietic stem cell transplantation, and therapeutic options for these infections are often complicated by associated toxicities. Genetically modified cytotoxic T-lymphocytes (CTLs) are designed to kill a specific virus that can cause infections. Depending on which virus a patient is infected with (ADV, BKV, CMV, JCV, or COVID-19), the CTLs will be designed to specifically attack that virus. Giving genetically modified CTLs may help to control the infection.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the feasibility and safety of administering genetically engineered glucocorticoid receptor knock out virus specific cytotoxic T-lymphocyte (CTL) lines in immunosuppressed cancer patients with viral infections (BKV, JCV, CMV, adenovirus, COVID19).

SECONDARY OBJECTIVES:

I. To obtain preliminary data about the efficacy of administering genetically engineered glucocorticoid receptor knock out virus specific CTL lines in immunosuppressed cancer patients with viral infections (BKV, JCV, CMV, adenovirus, COVID19).

II. To assess the persistence of the administered cells in the patients. III. To obtain data about relapse free survival (RFS) and overall survival (OS).

OUTLINE:

Patients receive virus-specific CTLs intravenously (IV) over 30 minutes. Patients with partial response, stable disease, or progressive disease may receive up to 8 additional infusions of virus-specific CTL at least 2 weeks between each infusion.

After completion of study treatment, patients are followed up yearly for 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients > or = 18 years of age or older.
* For BKV, ADV or CMV infections: Prior myeloablative or non-myeloablative allogeneic hematopoietic stem cell transplant using bone marrow, peripheral blood stem cells or single or double umbilical cord blood. For JC virus and COVID19 infection: no prior hematopoietic stem cell transplantation (HSCT) is required.
* For BKV infection, patients need to have polymerase chain reaction (PCR) positive for BKV (in peripheral blood or urine) with consistent clinical symptoms.
* For ADV infection, patients need to have PCR positive for ADV in peripheral blood AND/OR patients need to fit criteria of probable or definitive adenovirus organ disease.
* For CMV infection, patients need to have PCR positive for CMV in peripheral blood AND/OR patients need to fit criteria of probable or definitive CMV disease.
* For JCV, patients need to have documented JC viral encephalitis or JC end-organ disease.
* For COVID-19 infection, patients need to have COVID-19 related pneumonia/acute respiratory distress syndrome (ARDS) to be enrolled, defined as patients with a positive COVID-19 test (bronchoalveolar lavage [BAL], nasal or pharyngeal) and radiological and clinical signs of pneumonia or ARDS.
* Written informed consent from patient or designated power of attorney.
* Subjects are also are required to consent to PA17-0483 for long term follow up per the guidelines set forth by the Food and Drug Administrations' (FDA's) Biologic Response Modifiers Advisory Committee (BRMAC).
* Negative pregnancy blood test in female patients of childbearing potential, defined as not post-menopausal for 12 months or no previous surgical sterilization. Women of child bearing potential must be willing to use at least two forms of birth control during the study and for at least 6 months after stopping treatment. Acceptable forms of birth control include intrauterine device (IUD), hormonal methods (birth control pills, injections, and implants), condoms, diaphragms, tubal ligation, or vasectomy.

Exclusion Criteria:

* Patients who have received anti-thymocyte globulin (ATG) within 14 days or have received donor lymphocyte infusion (DLI) or campath within 28 days of enrollment.
* Patients with other uncontrolled infections (excluding human immunodeficiency virus [HIV]/acquired immunodeficiency syndrome [AIDS]). For bacterial infections, patients must be receiving definitive therapy and have signs of improving infection prior to enrollment as determined by the principal investigator (PI). For fungal infections, patients must be receiving definitive systemic anti-fungal therapy and have signs of improving infection prior to enrollment as determined by the PI.
* Patients with active steroid refractory graft versus host disease (GVHD).
* Patients on immunosuppressive therapy other than tacrolimus, sirolimus or steroids
* Active and uncontrolled relapse of malignancy. Patients with controlled malignancy on maintenance therapy would be eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-06 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of administering genetically engineered glucocorticoid receptor knock out virus specific cytotoxic T-lymphocyte (CTL) lines, as indicated by Overall Survival | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: May Daher, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org